CLINICAL TRIAL: NCT06023082
Title: A Single-Group Study to Examine the Efficacy of a Gut Health Supplement to Increase Metabolism, Improve Gut Health, and Support Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gut Health, UAB (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20349
Record Dates: First submitted 2023-08-28; First posted 2023-09-05 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Gut Health; Metabolism; Weight Loss; Energy
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Masking Description: Participants will be blinded to the brand and name of the supplement they are taking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colon Broom Premium supplement (Experimental): Participants will add 1 scoop (0.23 oz/ 6.47 g) to 12-14 fl oz of water, mix well and drink immediately. Participants will take the supplement 30 -60 minutes before their meal and will then drink an additional glass of water. Participants will be instructed not to take the supplement less than 2 hours before bedtime. The test product may be consumed before breakfast, lunch, or dinner.
  First week: Start with 1 serving per day Rest of the study period: Increase to 2 servings per day at 2 different times during the day.
  Interventions: Dietary Supplement: Colon Broom Premium supplement

INTERVENTIONS:
Dietary Supplement: Colon Broom Premium supplement — The product contains the following ingredients:
  Psyllium Seed Husk Powder L-Carnitine Tartrate Capsimax® Cayenne Fruit Extract Chromium (as Chromium Picolinate) Vitamin B6 (as Pyridoxine HCl) Vitamin B12 (as Cyanocobalamin) Iron

SUMMARY:
This study will evaluate the efficacy of Colon Broom Premium on gut health, metabolism, weight management, and energy levels. The study will be conducted as a virtual single-group trial in which all 120 participants will use the test product. This study will last 12 weeks, and participants will take the product daily. Participants will complete study-specific questionnaires at Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12. Participants will also provide body weight measurements and body circumference measurements at Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12.

Before & after photographs will be provided at Baseline and Week 12.

The Colon Broom Premium supplement contains psyllium seed husk powder, L-carnitine tartrate, CapsimaxⓇ cayenne fruit extract, chromium (as chromium picolinate), vitamin B6 (as pyridoxine HCl), vitamin B12 (as cyanocobalamin), and Iron.

The study Sponsor and product name will remain anonymous to participants throughout the trial. The Sponsor name or product name will not be included in any participant-facing documentation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between ages 30-50
* Have a BMI of 25 or more
* Have self-reported issues with gas, bloating, constipation, heartburn/acid reflux, abdominal pain, or digestion at least three times per week
* Be willing to maintain their standard dietary pattern, activity level, and body weight for the duration of the study
* Be generally healthy - do not live with any uncontrolled chronic disease

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* Anyone who is currently undergoing, or planning to to undergo any gut or weight-related procedures in the next 12 week.
* Anyone with a history of severe allergic reactions including but not limited to psyllium seed husk powder and strawberries
* Anyone taking any prescription medications targeting the gut
* Anyone taking any supplements targeting the gut in the past month
* Use of antibiotics in the past 3 months
* Women who are pregnant, breastfeeding, or attempting to become pregnant
* Anyone unwilling to follow the study protocol
* Anyone following any particular dietary regime, such as a ketogenic diet or intermittent fasting.
* Anyone who has had bariatric surgery in the past 6 months
* Anyone who has chronic constipation
* Anyone who has Irritable Bowel Disease (IBD)
* Anyone diagnosed with severe digestive issues

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Colon Broom Premium Supplement: Participants will add 1 scoop (0.23 oz/ 6.47 g) to 12-14 fl oz of water, mix well and drink immediately. Participants will take the supplement 30 -60 minutes before their meal and will then drink an additional glass of water. Participants will be instructed not to take the supplement less than 2 hours before bedtime. The test product may be consumed before breakfast, lunch, or dinner.
  First week: Start with 1 serving per day Rest of the study period: Increase to 2 servings per day at 2 different times during the day.
  Colon Broom Premium supplement: The product contains the following ingredients:
  Psyllium Seed Husk Powder L-Carnitine Tartrate Capsimax® Cayenne Fruit Extract Chromium (as Chromium Picolinate) Vitamin B6 (as Pyridoxine HCl) Vitamin B12 (as Cyanocobalamin) Iron
Period: Overall Study
Arm/Group | Colon Broom Premium Supplement
Started | 120
Completed | 98
Not Completed | 22
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 15
Not completed — Side effects | 5

BASELINE CHARACTERISTICS:
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.69 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87
  Black or African American | 15
  Hispanic or Latino | 7
  Asian | 3
  American Indian or Alaska Native | 1
  Mixed race | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 32.1535 (7.220633559)
Bodyweight [Mean (Standard Deviation); unit: Pounds (llbs)] | 198.0341667 (43.11105358)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Body Weight. [Baseline to Week 12]
Description: Participants will provide body weight measurements using a weighing scales.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: Pounds (lbs)
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
Pounds (lbs)
  Baseline | 194.81 (39.48)
  Week 1 | 194.35 (39.32)
  Week 2 | 194.17 (39.64)
  Week 3 | 193.68 (40.03)
  Week 4 | 192.84 (40.18)
  Week 6 | 192.81 (39.43)
  Week 8 | 192.18 (39.76)
  Week 10 | 191.19 (39.65)
  Week 12 | 189.86 (41.21)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

2. Primary Outcome: Changes in Waist Circumference. [Baseline to Week 12]
Description: Participants will independently measure their waist circumference in inches.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
Inches
  Baseline | 38.43 (6.30)
  Week 1 | 38.74 (5.76)
  Week 2 | 38.35 (5.61)
  Week 3 | 38.44 (5.97)
  Week 4 | 37.89 (5.87)
  Week 6 | 38.14 (5.46)
  Week 8 | 37.38 (6.17)
  Week 10 | 37.36 (6.10)
  Week 12 | 37.05 (5.82)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA

3. Primary Outcome: Changes in Hip Circumference. [Baseline to Week 12]
Description: Participants will independently measure their hip circumference in inches.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
Inches
  Baseline | 44.24 (6.34)
  Week 1 | 43.84 (5.85)
  Week 2 | 43.32 (5.64)
  Week 3 | 43.56 (5.79)
  Week 4 | 43.21 (5.71)
  Week 6 | 43.06 (6.02)
  Week 8 | 42.80 (5.98)
  Week 10 | 42.45 (6.61)
  Week 12 | 42.21 (6.15)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

4. Primary Outcome: Changes in Thigh Circumference. [Baseline to Week 12]
Description: Participants will independently measure their thigh circumference in inches.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
Inches
  Baseline | 25.12 (4.63)
  Week 1 | 24.84 (4.36)
  Week 2 | 24.79 (4.03)
  Week 3 | 24.36 (3.31)
  Week 4 | 24.68 (4.12)
  Week 6 | 24.37 (4.19)
  Week 8 | 24.13 (3.91)
  Week 10 | 23.80 (4.12)
  Week 12 | 24.03 (3.94)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

5. Secondary Outcome: Changes in Overall Health. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-perceived changes in overall health. On the scale, 1=worst response, and 5= the most favorable response.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.75 (0.77)
  Week 1 | 3.86 (0.66)
  Week 2 | 3.85 (0.68)
  Week 3 | 3.90 (0.72)
  Week 4 | 3.89 (0.68)
  Week 6 | 3.89 (0.65)
  Week 8 | 3.74 (0.81)
  Week 10 | 3.95 (0.67)
  Week 12 | 3.91 (0.85)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p = 0.4907, ANOVA — Baseline to Week 12 comparison

6. Secondary Outcome: Changes in Energy Levels. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-perceived changes in energy levels. On the scale, 1=worst response, and 5= the most favorable response.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 2.47 (0.68)
  Week 1 | 3.01 (0.64)
  Week 2 | 3.05 (0.65)
  Week 3 | 3.11 (0.71)
  Week 4 | 3.15 (0.68)
  Week 6 | 3.16 (0.81)
  Week 8 | 3.13 (0.91)
  Week 10 | 3.18 (0.77)
  Week 12 | 3.22 (0.87)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

7. Secondary Outcome: Changes in Tiredness. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-perceived changes in tiredness. On the scale, 1=worst response, and 5= the most favorable response.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 1.80 (0.72)
  Week 1 | 2.52 (0.98)
  Week 2 | 2.52 (0.99)
  Week 3 | 2.75 (1.05)
  Week 4 | 2.67 (1.12)
  Week 6 | 2.71 (1.08)
  Week 8 | 2.69 (1.11)
  Week 10 | 2.70 (1.18)
  Week 12 | 2.90 (1.07)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

8. Secondary Outcome: Changes in Overall Mood. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-perceived changes in overall mood. On the scale, 1=worst response, and 5= the most favorable response.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.30 (0.68)
  Week 1 | 3.75 (0.62)
  Week 2 | 3.74 (0.67)
  Week 3 | 3.69 (0.65)
  Week 4 | 3.75 (0.68)
  Week 6 | 3.71 (0.74)
  Week 8 | 3.69 (0.81)
  Week 10 | 3.77 (0.77)
  Week 12 | 3.80 (0.75)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

9. Secondary Outcome: Changes in Mental Wellbeing. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-perceived changes in mental wellbeing. On the scale, 1=worst response, and 5= the most favorable response.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.47 (0.71)
  Week 1 | 3.81 (0.62)
  Week 2 | 3.81 (0.60)
  Week 3 | 3.78 (0.71)
  Week 4 | 3.78 (0.71)
  Week 6 | 3.80 (0.80)
  Week 8 | 3.67 (0.79)
  Week 10 | 3.82 (0.73)
  Week 12 | 3.84 (0.80)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p = 0.0016, ANOVA — Baseline to Week 12 comparison

10. Secondary Outcome: Changes in Ability to Focus. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-perceived changes in ability to focus. On the scale, 1=worst response, and 5= the most favorable response.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.11 (0.93)
  Week 1 | 3.55 (0.79)
  Week 2 | 3.65 (0.79)
  Week 3 | 3.68 (0.72)
  Week 4 | 3.66 (0.86)
  Week 6 | 3.63 (0.92)
  Week 8 | 3.59 (0.85)
  Week 10 | 3.69 (0.82)
  Week 12 | 3.77 (0.89)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

11. Secondary Outcome: Changes in Amount of Daily Leisure Time Spent Doing Something Active. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-reported changes in the amount of daily leisure time spent active. On the scale, 1=least amount of time, and 5= the most amount of time. 1= 0-15min; 2= 15-30min; 3= 30-60min; 4=60-90 min; 5=more than 90min
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 2.61 (1.08)
  Week 1 | 3.04 (1.15)
  Week 2 | 3.08 (1.07)
  Week 3 | 3.23 (1.17)
  Week 4 | 3.11 (1.10)
  Week 6 | 3.13 (1.18)
  Week 8 | 3.05 (1.16)
  Week 10 | 3.15 (1.14)
  Week 12 | 3.21 (1.21)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

12. Secondary Outcome: Changes in Frequency of Constipation. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-reported changes in frequency of constipation. On the scale, 1=worst response, and 5= the most favorable response. 1= Never; 2= Less than once per week; 3= Once per week; 4= 2-5 times per week; 5= More than 5 times per week.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.01 (1.02)
  Week 1 | 3.64 (1.20)
  Week 2 | 3.94 (1.03)
  Week 3 | 3.95 (1.16)
  Week 4 | 4.01 (1.10)
  Week 6 | 3.98 (1.19)
  Week 8 | 3.91 (1.18)
  Week 10 | 3.99 (1.14)
  Week 12 | 4.10 (1.12)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

13. Secondary Outcome: Changes in Severity of Constipation. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-reported changes in severity of constipation. On the scale, 1=worst response, and 5= the most favorable response. 1= Not noticeable; 2= Barely noticeable; 3= Moderate; 4= Distracting ; 5= Severe.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.34 (0.90)
  Week 1 | 3.70 (0.82)
  Week 2 | 3.89 (0.87)
  Week 3 | 3.96 (0.92)
  Week 4 | 3.97 (0.94)
  Week 6 | 4.06 (0.91)
  Week 8 | 3.81 (0.98)
  Week 10 | 3.88 (0.93)
  Week 12 | 4.34 (0.87)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p = 0.0002, ANOVA — Baseline to Week 12 comparison

14. Secondary Outcome: Changes in Bowel Movement Regularity. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-reported changes in bowel movement regularity. On the scale, 1=worst response, and 5= the most favorable response. 1= Never; 2= Less than once per week; 3= Once per week; 4= 2-5 times per week; 5= More than 5 times per week.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.94 (0.84)
  Week 1 | 4.34 (0.71)
  Week 2 | 4.28 (0.75)
  Week 3 | 4.39 (0.67)
  Week 4 | 4.34 (0.88)
  Week 6 | 4.46 (0.71)
  Week 8 | 4.41 (0.67)
  Week 10 | 4.15 (1.03)
  Week 12 | 4.31 (0.90)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p = 0.001, ANOVA — Baseline to Week 12 comparison

15. Secondary Outcome: Changes in Frequency of Gas. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-reported changes in frequency of gas. On the scale, 1=worst response, and 5= the most favorable response. 5= Never; 4= Less than once per week; 3= Once per week; 2= 2-5 times per week; 1= More than 5 times per week.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 1.71 (0.68)
  Week 1 | 2.32 (1.10)
  Week 2 | 2.63 (1.20)
  Week 3 | 2.73 (1.20)
  Week 4 | 2.93 (1.20)
  Week 6 | 2.93 (1.27)
  Week 8 | 3.00 (1.24)
  Week 10 | 3.11 (1.26)
  Week 12 | 3.16 (1.25)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

16. Secondary Outcome: Changes in Severity of Gas. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-reported changes in severity of gas. On the scale, 1=worst response, and 5= the most favorable response. 5= Not noticeable; 4= Barely noticeable; 3= Moderate; 2= Distracting; 1= Severe.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 2.76 (0.69)
  Week 1 | 3.35 (0.88)
  Week 2 | 3.58 (0.89)
  Week 3 | 3.64 (0.95)
  Week 4 | 3.82 (0.86)
  Week 6 | 3.84 (0.90)
  Week 8 | 3.74 (0.97)
  Week 10 | 3.82 (0.92)
  Week 12 | 3.92 (0.91)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

17. Secondary Outcome: Changes in Frequency of Bloating. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-reported changes in frequency of bloating. On the scale, 1=worst response, and 5= the most favorable response. 5= Never; 4= Less than once per week; 3= Once per week; 2= 2-5 times per week; 1= More than 5 times per week.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 2.13 (0.94)
  Week 1 | 2.71 (1.20)
  Week 2 | 3.16 (1.23)
  Week 3 | 3.22 (1.22)
  Week 4 | 3.41 (1.20)
  Week 6 | 3.52 (1.21)
  Week 8 | 3.50 (1.20)
  week 10 | 3.66 (1.26)
  Week 12 | 3.66 (1.20)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

18. Secondary Outcome: Changes in Severity of Bloating. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-reported changes in severity of bloating. On the scale, 1=worst response, and 5= the most favorable response. 5= Not noticeable; 4= Barely noticeable; 3= Moderate; 2= Distracting; 1= Severe.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 2.75 (0.88)
  Week 1 | 3.47 (0.95)
  Week 2 | 3.74 (0.92)
  Week 3 | 3.73 (0.99)
  Week 4 | 3.79 (1.03)
  Week 6 | 3.97 (0.93)
  Week 8 | 3.84 (0.96)
  Week 10 | 3.92 (1.02)
  Week 12 | 4.03 (0.86)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Baseline to Week 12 comparison; Test type: Other; p < 0.0001, ANOVA

19. Secondary Outcome: Changes in Discomfort Associated With Gut Issues. [Baseline to Week 12]
Description: Survey-based assessment on a 7-point Likert scale of participant-reported changes in frequency of constipation. On the scale, 1=worst response, and 7= the most favorable response. 7= No discomfort at all; 6= Minor discomfort; 5= Mild discomfort; 4= Moderate discomfort; 3= Moderately severe discomfort; 2= Severe discomfort; 1= Very severe discomfort.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, and Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 3.86 (1.11)
  Week 1 | 5.27 (1.14)
  Week 2 | 5.52 (1.14)
  Week 3 | 5.64 (1.26)
  Week 4 | 5.58 (1.30)
  Week 6 | 5.71 (1.26)
  Week 8 | 5.82 (1.11)
  Week 10 | 5.72 (1.30)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 10 comparison

20. Secondary Outcome: Changes in Frequency of Feeling Hunger After Eating a Meal. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-report changes in frequency of feeling hungry even after eating a meal. On the scale, 1=worst response, and 5= the most favorable response. 5= Never; 4= Less than once per week; 3= Once per week; 2= 2-5 times per week; 1= More than 5 times per week.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 2.54 (1.10)
  Week 1 | 3.38 (1.24)
  Week 2 | 3.69 (1.24)
  Week 3 | 3.71 (1.17)
  Week 4 | 3.71 (1.09)
  Week 6 | 3.78 (1.17)
  Week 8 | 3.81 (1.20)
  Week 10 | 3.80 (1.07)
  Week 12 | 3.86 (1.16)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

21. Secondary Outcome: Changes in Number of Bowel Movements Per Week. [Baseline to Week 12]
Description: Participants were asked to report the number of bowel movements they had in the previous week.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: Number of bowel movements per week
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
Number of bowel movements per week
  Baseline | 5.63 (3.96)
  Week 1 | 7.13 (4.15)
  Week 2 | 7.19 (4.51)
  Week 3 | 7.26 (4.05)
  Week 4 | 7.75 (4.71)
  Week 6 | 7.59 (4.52)
  Week 8 | 7.21 (4.68)
  Week 10 | 7.41 (4.48)
  Week 12 | 7.21 (4.10)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

22. Secondary Outcome: Changes in the Frequency of Experiencing Food Cravings. [Baseline to Week 12]
Description: Survey-based assessment on a 5-point Likert scale of participant-reported changes in frequency of constipation. On the scale, 1=worst response, and 5= the most favorable response. 5= Never; 4= Less than once per week; 3= Once per week; 2= 2-5 times per week; 1= More than 5 times per week.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 1.94 (0.97)
  Week 1 | 2.77 (1.23)
  Week 2 | 2.95 (1.17)
  Week 3 | 3.16 (1.13)
  Week 4 | 3.27 (1.15)
  Week 6 | 3.23 (1.24)
  Week 8 | 3.28 (1.23)
  Week 10 | 3.42 (1.25)
  Week 12 | 3.47 (1.24)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

23. Secondary Outcome: Changes in Frequency of Overeating. [Baseline to Week 12]
Description: as for outcome 22
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8, Week 10, and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Colon Broom Premium Supplement
Number analyzed (Participants) | 98
score on a scale
  Baseline | 2.47 (1.14)
  Week 1 | 3.35 (1.19)
  Week 2 | 3.60 (1.13)
  Week 3 | 3.53 (1.20)
  Week 4 | 3.71 (1.15)
  Week 6 | 3.64 (1.24)
  Week 8 | 3.70 (1.22)
  Week 10 | 3.74 (1.20)
  Week 12 | 3.75 (1.16)
Statistical Analysis 1: Comparison: Colon Broom Premium Supplement; Test type: Other; p < 0.0001, ANOVA — Baseline to Week 12 comparison

24. Other Pre Specified Outcome: Visual Changes in Weight. [Baseline to Week 12]
Description: At baseline and endline, participants provided three photos from their chin down to their knees at the following angles: front-facing, side profile, and facing backward. These photos were not analyzed or included in the data analysis.
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 12-week study period.
Arm/Group | Colon Broom Premium Supplement
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 5/120
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Colon Broom Premium Supplement (N=120)
Diarrhea (Gastrointestinal disorders) | 4
Bloating and Gas (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
Reliance on self-reported data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT06023082/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT06023082/ICF_001.pdf